CLINICAL TRIAL: NCT05237713
Title: A Phase II, Single-Arm, Open-Label Study to Assess the Efficacy and Safety of Canakinumab for the Treatment of Anemia in Patients With IPSS-R Very Low, Low, or Intermediate Risk Myelodysplastic Syndromes or MDS/MPN
Brief Title: Efficacy and Safety of Canakinumab for the Treatment of Anemia in LR-MDS Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment. It is not considered likely that the CANFIRE trial will be able to reach the target number of patients. Clinical responders will be further treated within the trial (expected duration: 3 years after stop of enrollment).
Sponsor: University of Leipzig (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Anne Sophie Kubasch, Coordinating Investigator, University of Leipzig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CANFIRE
Record Dates: First submitted 2022-01-21; First posted 2022-02-14 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Anemia; Myelodysplastic Syndromes
Keywords: anemia; low risk MDS; inflammation; IL-1beta blockade; NLRP3 activation
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes; Inflammation | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Canakinumab treatment (Other): 200 mg canakinumab subcutaneously every three weeks
  Interventions: Drug: Canakinumab Injection

INTERVENTIONS:
Drug: Canakinumab Injection — Administration for a duration of 6 months for all patients and in case of response further treatment for up to three years
  Other Names: Ilaris(R)

SUMMARY:
Hematologic improvement of erythrocytes after 6 months of canakinumab treatment.

DETAILED DESCRIPTION:
To study the erythroid response rate (HI-E) of canakinumab in patients with IPSS-R very low, low, or intermediate risk MDS or MDS/MPN after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of

   1. Lower-risk myelodysplastic syndrome (MDS) OR
   2. Myelodysplastic/myeloproliferative neoplasm (MDS/MPN) including MDS/MPN-RS-T, MDS/MPNu, aCML, or CMML (as per the World Health Organization [WHO] 2016 classification) Note: Diagnoses will be confirmed by central morphological review during screening assessment
2. Very low, low or intermediate risk disease MDS with up to 3.5 points according to the revised International Prognostic Scoring System (IPSS-R) classification (to be confirmed during screening assessment). For MDS/MPN < 10% bone marrow blasts at screening. For CMML low or intermediate risk according to CMML-Specific Prognostic Scoring System (CPSS Score).
3. Symptomatic anemia (all NTD, LTB, or HTB): has to be documented in the 16 weeksbaseline period ending on the day of inclusion. Patients should be registered only if it is expected at time of registration that

   1. a valid and complete hemoglobin and transfusion history will be available at inclusion AND
   2. the hemoglobin mean over the baseline period will be less than 10 g/dL OR three or more RBC-transfusions will have been given during the baseline period documenting transfusion dependence.
4. Documented transfusion strategy: A transfusion trigger threshold is needed which characterizes the transfusion strategy - ideally for the whole baseline period, but at least for the time from registration to the end of the study.
5. Relapsed / refractory / intolerant / ineligible (endogenous serum erythropoietin levels ≥ 200 U/L) to ESA treatment
6. Age ≥ 18 years
7. Written informed consent

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the trial.

Compliance with major study procedures

1. Patient does not accept bone marrow sampling during screening and treatment period.
2. Patient does not accept peripheral blood sampling for screening and during treatment.
3. Patient does not accept subcutaneous application of canakinumab every three weeks

   Contraindications
4. Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding

   a. iron deficiency must be determined by calculated transferrin saturation (iron/total iron binding capacity) ≤ 20%, or serum ferritin ≤ 15 µg/L
5. Prior allogeneic or autologous stem cell transplant
6. Known history of diagnosis of AML

   Safety
7. Severe neutropenia defined by ANC ≤ 0.5 Gpt/l
8. Severe thrombocytopenia with platelets (PLT) < 30 Gpt/L
9. Serum creatinine > 1.5x ULN OR measured or calculated creatinine clearance < 40 ml/min (NOTE: creatinine clearance should be calculated per institutional standard. GFR can also be used)
10. Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) or alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT) ≥ 3.0 x upper limit of normal (ULN) - both have to be measured
11. Eastern Cooperative Oncology Group (ECOG) > 2
12. Total bilirubin ≥ 2.0 x ULN

    1. higher levels are acceptable if these can be attributed to active red blood cell precursor destruction within the bone marrow (ie, ineffective erythropoiesis).
    2. subjects are excluded if there is evidence of autoimmune hemolytic anemia manifested as a corrected reticulocyte count of > 2% with either a positive Coombs' test or over 50% indirect bilirubin
13. Active second malignancy at time of study entry
14. Prior history of malignancies, other than MDS, unless the subject has been free of the disease for ≥ 5 years. However, subjects with the following history/concurrent conditions are allowed:

    1. Basal or squamous cell carcinoma of the skin
    2. Carcinoma in situ of the cervix
    3. Carcinoma in situ of the breast
    4. Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system)
15. Major surgery within 8 weeks prior to screening (NOTE: Subjects must have completely recovered from any previous surgery prior to inclusion)
16. Myocardial infarction, uncontrolled angina, uncontrolled heart failure, or uncontrolled cardiac arrhythmia within 6 months prior to screening
17. Positive test result as an indicator for active or latent tuberculosis (evaluation performed per local treatment guidelines or clinical practice)
18. Subjects with suspected or proven immunocompromised state or infections, including:

    1. Known history of testing positive for Human Immunodeficiency Virus (HIV) infections.
    2. Known active or recurrent, hepatitis B and C (positive or indeterminate laboratory results).
    3. Those with any other medical condition such as active infection, treated or untreated, which in the opinion of the investigator places the subject at an unacceptable risk for participation in immunomodulatory therapy.
    4. Those requiring systemic or local treatment with any immune modulating agent in doses with systemic effects e.g.: Prednisone >20 mg (or equivalent) oral or intravenous daily for >14 days; Prednisone > 5 mg and ≤ 20 mg (or equivalent) daily for > 30 days; Equivalent dose of methotrexate >15 mg weekly.
    5. History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational product (see Investigator´s Brochure).

    Excluded treatments before and during study treatment
19. Anticancer cytotoxic chemotherapeutic agent or treatment for at least 14 days prior to registration and during study treatment
20. Corticosteroids or other immunosuppressive therapies (TNF-Blocker, other IL-1 Blocking Agent, Disease-modifying anti-rheumatic drugs (DMARDs) including ciclosporin, cyclophosphamide, hydroxychloroquine, leflunomide, methotrexate, mycophenolate, sulfasalazine) for at least 14 days prior to registration and during study treatment
21. Treatment with ESAs, luspatercept, granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF) for at least 14 days prior to registration and during study treatment
22. Treatment with disease modifying agents (eg, immune-modulatory drugs [IMiDs such as lenalidomide, hypomethylating agents] or experimental agents for underlying MDS disease for at least 14 days prior to registration and during study treatment
23. Prior treatment with canakinumab
24. Live vaccination during study treatment

    Special considerations for females
25. Pregnant or breastfeeding females
26. Positive pregnancy test in women of childbearing potential NOTE: Urine or serum pregnancy test should be repeated within 3 days prior to receiving study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test is required additionally
27. Female subjects of childbearing potential unwilling to use an adequate method of contraception for the course of the study through 90 days after the last dose of study medication NOTE: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

    Special considerations for males
28. Male subjects with procreative capacity not willing to use an adequate method of contraception, starting with the first dose of study therapy through 90 days after the last dose of study therapy NOTE: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

    Regulatory requirements
29. Participation in other interventional trials
30. Patients under legal supervision or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
HI-E after 6 months of treatment | 6 months
  Erythroid response rate (HI-E) of canakinumab

SECONDARY OUTCOMES:
HI-E response duration | up to three years
  Duration of erythroid response rate will be measured up to loss of response or reaching end of study (after max. 3 years of treatment)
Number of (serious) adverse events | up to three years
  The safety profile of canakinumab will be described by collecting AE (adverse event) and SAE (serious adverse event) information up to the start of new treatment or reaching end of study (after max. 3 years of treatment). Special consideration will be laid on events that lead to treatment discontinuation.
Disease progression | after 24 weeks
  Proportion of disease progression (after reaching PD at any time during the trial after primary end-point visit)
Impact of canakinumab on quality of life by using the validated Quality of Life in Myelodysplasia Scale (QUALMS) | From the date of treatment start until the end of study, assessed up to 36 months
  QoL assessment using the QUALMS questionnaire up to end of treatment:
  38-item assessment tool for patients with Myelodysplastic Syndromes (MDS) QUALMS scores ranged from 24 to 99, with higher scores for better outcome
Impact of canakinumab on quality of life by using the validated European Organisation for Research and Treatment of Cancer Core Quality of Life questionnaire (EORTC QLQ-C30) | From the date of treatment start until the end of study, assessed up to 36 months
  QoL assessment using the EORTC-C30 questionnaire up to end of treatment:
  To assess patient-reported quality of life during canakinumab treatment: 30 questions assessing the quality of life of oncology patients across 10 subscales will be analyzed. All subscales have a score range from 0 to 100 points.
  Function subscales: a higher score represents a higher quality of life. Symptoms subscales: higher score represents higher level of symptoms/problems, i.e., represents lower quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sophie Kubasch, Dr., Principal Investigator — University Leipzig
Locations (3):
- Germany (3):
  - Medizinisches Versorgungszentrum "Onkologischer Schwerpunkt am Oskar- Helene-Heim", Berlin
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden Medizinischen Klinik und Poliklinik I / Hämatologie, Dresden
  - Klinik und Poliklinik für Hämatologie und Zelltherapie, Hämostaseologie, Leipzig

IPD SHARING:
Plan to Share IPD: No